CLINICAL TRIAL: NCT03474757
Title: Treatment Pattern of NOACs (Non-vitamin K Oral Anticoagulants) in Outpatient Users in Colombian Databases - TREND Colombia
Brief Title: Treatment Pattern of NOACs (Non-vitamin K Oral Anticoagulants) in Outpatient Users in Colombian Databases
Acronym: TREND
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20104
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SPAF patients in Colombia_Rivaroxaban: First time users of rivaroxaban in the Audifarma database
  Interventions: Other: Data Collection
- SPAF patients in Colombia_Dabigatran: First time users of dabigatran in the Audifarma database
  Interventions: Other: Data Collection
- SPAF patients in Colombia_Apixaban: First time users of apixaban in the Audifarma database
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Data will be extracted from July 2009 to the last available database extraction

SUMMARY:
This population-based descriptive study will characterize first-time users of three NOACs (rivaroxaban, dabigatran and apixaban) in prevention of stroke in non-valvular atrial fibrillation (SPAF) patients and will assess the patterns of drug utilization in routine general practice in Colombia

ELIGIBILITY:
Inclusion Criteria:

* First prescription of NOACs (rivaroxaban, dabigatran and apixaban) in the outpatient setting.
* Non valvular Atrial Fibrillation (NVAF) Patients
* aged ≥18 years
* at least one year of enrollment in the Audifarma database
* one year since first encounter with healthcare provider will be included in the study

Exclusion Criteria:

* Patients with any record of index drug prescription prior to the enrolment period.
* Patients who qualify as members of more than one cohort study on the same day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the population from the Audifarma database, the study will be comprised of three separate cohorts of first time users of rivaroxaban, dabigatran and apixaban using the first prescription date (index date) of the respective drug (index drug). All patients aged ≥18 years with at least one year of enrollment in the databases and one year since first encounter with healthcare provider will be included in the study.
Sampling Method: Probability Sample
Enrollment: 10528 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Age | At Baseline
Sex | At Baseline
Co-morbidity | At Baseline
Healthcare utilization | Up to 2 years
  Primary Care Physicians visits, Outpatient visits and Hospital admissions
Proportion of Naive to non-naive patient | At Baseline
Dose at first prescription | Up to 6 years
Duration of treatment | Up to 6 years
Discontinuation | Up to 6 years
Switch to another study drug | Up to 6 years

SECONDARY OUTCOMES:
Time trends of usage of study medications | Up to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Colombia

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=20104&attachmentIdentifier=56598450-2870-4624-96d2-d9e0bbaf1111&fileName=20104_study_synopsis_revised_2020-03-25.pdf&versionIdentifier=